CLINICAL TRIAL: NCT03186937
Title: A Window of Opportunity Study of Methionine Deprivation in Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding and slow enrollment
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Avon Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UW16083; 2016-1532 (Other: Institutional Review Board); NCI-2017-01047 (Registry Identifier: NCI CTRP); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 11/23/2020 (Other: UW Madison)
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hominex-2 (Experimental): Participants will receive an individualized dietary prescription that incorporates a methionine-free amino acid-modified medical food (Hominex-2, Abbott Nutrition) supplemented with low-methionine foods. Hominex-2 contains a mixture of L-amino acids but lacks methionine.
  Participants will be asked to have an optional non-contrast MRI to assess body composition prior to and at completion of the methionine-restricted (MR) diet. Not completing a scheduled MRI is not considered a protocol deviation.
  Participants will be followed for 30 days after surgery or biopsy date. Subjects removed from study for unacceptable adverse events (AEs) will be followed until resolution or stabilization of the AE.
  Interventions: Dietary Supplement: hominex-2

INTERVENTIONS:
Dietary Supplement: hominex-2 — Hominex-2 is a methionine-free amino acid modified medical supplement
  Other Names: Nut.Tx; Metabol; Methio-Fr

SUMMARY:
Given preliminary data demonstrating that methionine deprivation enhances cell surface expression of TRAIL receptor-2, the objective of this clinical trial is to confirm that methionine restriction enhances its expression in triple negative breast cancer and to establish the feasibility and acceptability of this dietary intervention in humans. This study will also examine the effect of methionine restriction on cancer stem cells and metabolic health.

DETAILED DESCRIPTION:
Under the supervision of a registered dietitian, subjects will receive an individualized dietary prescription that incorporates a methionine-free amino acid-modified medical food (Hominex-2, Abbott Nutrition) supplemented with low-methionine foods. Hominex-2 contains a mixture of L-amino acids but lacks methionine. Subjects will be instructed in the preparation of Hominex-2 beverages (approximately 4-5 per day or per dietician recommendation) to deliver 100% of daily protein requirements (0.8 g/kg/day) and 40-45% of the caloric requirements. The remaining calories will be met with low-methionine foods, including fruits, vegetables, grains (e.g., specified cereal and bread), margarine and cooking oils. Subjects will be provided with a list of foods that are low in methionine. Calories will not be restricted. Subjects will be encouraged to follow their usual level of physical activity and instructed to maintain a daily diet and exercise diary that will be reviewed weekly by the dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed operable triple negative breast cancer

  * ER (estrogen receptors) and PR (progesterone receptors) expression must be < 2%
  * HER2 must negative as shown be either 0 or 1+ by immunohistochemistry (if 2+, in situ hybridization method used to define HER2) OR by a HER2: 17 centromere signal of <2.0 using a standard in situ hybridization method.
* No prior therapy for current breast cancer
* Operable breast cancer. Participants who are planned to undergo neo-adjuvant chemotherapy are eligible as long as they consent to an additional breast biopsy following the dietary intervention immediately prior to starting chemotherapy
* ECOG (Eastern Cooperative Oncology Group) performance status ≤1
* Ability to understand and the willingness to sign a written informed consent document
* Serum creatinine <ULN (upper limit of normal)
* Non-pregnant. Women of childbearing potential must have a negative pregnancy test to participate in this study
* Women of childbearing potential must agree to use effective contraceptives (as discussed with their physician) while participating in this study

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients not able to swallow oral medications or with gastrointestinal conditions that may impact absorption of oral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change in cell surface expression of TRAIL receptor-2 | Up to 3 weeks
  To determine if methionine restriction can enhance the cell surface expression of TRAIL receptor-2 in triple negative breast cancers.

SECONDARY OUTCOMES:
Safety and tolerability of methionine measured by number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 3 weeks
  To examine the safety and tolerability of methionine restriction in participants with operable triple-negative breast cancer, measured by the number of participants with treatment-related adverse events as assessed by CTCAE v4.0.
Effect of methionine restriction on cancer stem cell markers CD44 and CD24 | Up to 3 weeks
  To examine the effect of methionine restriction on the expression of the cancer stem cell markers CD44 and CD24 by immunohistochemistry. Five to ten slides from each time point will be evaluated from baseline and after completion of the methionine restricted diet.
Change in plasma concentrations | Up to 3 weeks
  To evaluate plasma concentrations of methionine and methionine metabolites before and after methionine restriction. Blood will be collected after an overnight fast before dietary methionine restriction, weekly during methionine restriction and at the completion of the diet. Plasma concentration will be determined by high-throughput targeted LC-MS (liquid chromatography--mass spectrometry) assay.
Change in subject weight | Up to 3 weeks
  To evaluate subject weight before and after dietary methionine restriction. Subjects will be weighed before starting the diet and weekly (every 7 days +/- 1).
Change in subject BMI | Up to 3 weeks
  To evaluate subject BMI before and after dietary methionine restriction. Subjects will be weighed before starting the diet and weekly (every 7 days +/- 1).
Change in subject waist circumference | Up to 3 weeks
  To evaluate subject BMI, waist circumference and metabolic indices before and after dietary methionine restriction. Waist circumference will be measured before starting the diet and weekly (every 7 days +/- 1) while on the methionine restricted diet.
Change in subject metabolic indices | Up to 3 weeks
  To evaluate subject metabolic indices before and after dietary methionine restriction.
Change in body composition | Up to 3 weeks
  To evaluate body composition before and after dietary methionine restriction

CONTACTS AND LOCATIONS:
Overall Officials: Kari Wisinski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UW Carbone Cancer Center Homepage — http://www.uwhealth.org/uw-carbone-cancer-center/47424